CLINICAL TRIAL: NCT03052608
Title: A PHASE 3, RANDOMIZED, OPEN-LABEL STUDY OF LORLATINIB (PF-06463922) MONOTHERAPY VERSUS CRIZOTINIB MONOTHERAPY IN THE FIRST-LINE TREATMENT OF PATIENTS WITH ADVANCED ALK-POSITIVE NON-SMALL CELL LUNG CANCER
Brief Title: A Study Of Lorlatinib Versus Crizotinib In First Line Treatment Of Patients With ALK-Positive NSCLC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B7461006; 2023-509169-19-00 (Registry Identifier: CTIS (EU))
Expanded Access: NCT03127618 (Approved for marketing)
Record Dates: First submitted 2017-01-20; First posted 2017-02-14 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: ALK; anaplastic lymphoma kinase; Non-Small-Cell Lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lorlatinib; Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lorlatinib (Experimental): Lorlatinib single agent, 100 mg (4 x 25 mg) oral tables, QD, continuously
  Interventions: Drug: Lorlatinib
- Crizotinib (Active Comparator): Crizotinib single agent, 250 mg (1 x 250) oral capsules, BID, continuously
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Lorlatinib — ALK-positive NSCL treatment
  Other Names: PF-06463922
  Arms: Lorlatinib
Drug: Crizotinib — ALK-positive NSCL treatment
  Other Names: Xalkori
  Arms: Crizotinib

SUMMARY:
A phase 3 study to demonstrate whether lorlatinib given as monotherapy is superior to crizotinib alone in prolonging the progression-free survival in advanced ALK-positive NSCLC patients who are treatment naïve and to compare lorlatinib to crizotinib with respect to overall survival in the same population

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of locally advanced or metastatic ALK-positive NSCLC; at least 1 extracranial measurable target lesion not previously irradiated. CNS metastases allowed if asymptomatic and not currently requiring corticosteroid treatment.
* Availability of an archival FFPE tissue specimen.
* No prior systemic NSCLC treatment.
* ECOG PS 0, 1, or 2.
* Age ≥18 years .
* Adequate Bone Marrow, Liver, Renal, Pancreatic Function
* Negative pregnancy test for females of childbearing potential

Exclusion Criteria:

* Spinal cord compression unless good pain control attained
* Major surgery within 4 weeks prior to randomization.
* Radiation therapy within 2 weeks prior to randomization, including stereotactic or partial brain irradiation. Whole brain irradiation within 4 weeks prior to randomization
* Active bacterial, fungal, or viral infection
* Clinically significant cardiovascular disease, active or within 3 months prior to enrollment. Ongoing cardiac dysrhythmias, uncontrolled atrial fibrillation, bradycardia or congenital long QT syndrome
* Predisposing characteristics for acute pancreatitis in the last month prior to randomization.
* History of extensive, disseminated, bilateral or presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease
* Active malignancy (other than NSCLC, non melanoma skin cancer, in situ cervical cancer, papillary thyroid cancer, LCIS/DCIS of the breast, or localized prostate cancer) within the last 3 years prior to randomization.
* Concurrent use of any of the following food or drugs within 12 days prior to the first dose of lorlatinib or crizotinib.

  1. known strong CYP3A inhibitors .
  2. known strong CYP3A inducers
  3. known P gp substrates with a narrow therapeutic index
* Concurrent use of CYP3A substrates with narrow therapeutic indices within 12 days prior to the first dose of lorlatinib or crizotinib.
* Other severe acute or chronic medical or psychiatric condition, including recent or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or interfere with the interpretation of study results
* Investigational site staff members directly involved in the conduct of the study and their family members, or Pfizer employees, including their family members, directly involved in the conduct of the study.
* Participation in other studies involving investigational drug(s) within 2 weeks prior to study entry and/or during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2028-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (161):
- United States (31):
  - Florida Cancer Specialists, Altamonte Springs, Florida
  - Florida Cancer Specialists, Brandon, Florida
  - Florida Cancer Specialists, Clearwater, Florida
  - Florida Cancer Specialists, Gainesville, Florida
  - Florida Cancer Specialists, Largo, Florida
  - Florida Cancer Specialists, Lecanto, Florida
  - Florida Cancer Specialists, Orange City, Florida
  - Florida Cancer Specialists, Orlando, Florida
  - Florida Cancer Specialists, Spring Hill, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, Tampa, Florida
  - Florida Cancer Specialists, Tavares, Florida
  - Florida Cancer Specialists, The Villages, Florida
  - Florida Cancer Specialists, Winter Park, Florida
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ophthalmic Consultants of Boston Inc, Boston, Massachusetts
  - The William P. Beetham Eye Institute, Joslin Diabetes Center, Boston, Massachusetts
  - University of Rochester Cancer Center Pharmacy, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute., Nashville, Tennessee
  - Tennessee Oncology, PLLC, Shelbyville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - University of Washington Medical Center, Seattle, Washington
- Argentina (2):
  - Centro de Investigacion Pergamino SA, Pergamino, Buenos Aires
  - Centro Medico Austral, CABA
- Australia (4):
  - Bendigo Day Surgery Collection Centre and Laboratory, Bendigo, Victoria
  - Bendigo Medical Imaging, Bendigo Hospital, Bendigo, Victoria
  - Melbourne Pathology, Bendigo, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Grand Hopital de Charleroi - Site Notre Dame, Charleroi, Belgium
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- China (8):
  - The Affiliated Hospital of Military Medical Sciences, Beijing, Beijing Municipality
  - Jilin Provincial Cancer Hospital, Changchun, Jilin
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Department of Respiratory,the First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Guangdong General Hospital, Guangzhou
- Czechia (2):
  - Fakultni nemocnice Olomouc, Klinika plicnich nemoci a tuberkulozy, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (16):
  - Hopital Haut-Léveque-Centre François Magendie, Pessac, Aquitaine
  - Hopital de Chevilly Larue, Chevilly-Larue
  - Centre Hospitalier du Mans, Le Mans
  - Institut Paoli-Calmettes, Marseille
  - Département d'Imagerie Médicale, Marseille
  - Hôpital Nord, Marseille
  - Service Ophtalmologie, Marseille
  - Groupe Hospitalier Bichat Claude Bernard, AP-HP, Paris
  - CHU de Rennes Hopital Pontchaillou, Rennes
  - CHU de Rennes, Hopital Pontchaillou, Rennes
  - Hopital Foch, Suresnes
  - Hopital Larrey, Toulouse
  - Hopital Pierre Paul Riquet, Toulouse
  - Hôpital Larrey, Toulouse
  - Department d'imagerie medicale, Villejuif
  - Institut Gustave Roussy, Villejuif
- Germany (8):
  - Uberortliche Radiologische Gemeinschaftspraxis Dr. med. Marc Amler, Dresden
  - Technische Universitat Dresden , Medizinische Fakultat Carl Gustav Carus, Dresden
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Universitatsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Innere Medizin V, Homburg - Saar
  - Universitätsklinikum des Saarlandes, Homburg - Saar
  - Universitatsklinikum Regensburg, Institut fur Rontgendiagnostik, Regensburg
  - Universitatsklinikum Regensburg, Klinik und Poliklinik fur Innere Medizin II, Regensburg
- Hong Kong (3):
  - The University of Hong Kong, Department of Clinical Oncology, Hong Kong
  - The University of Hong Kong, Department of Medicine, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- India (5):
  - Artemis Hospital, Gurugram, Haryana
  - Manipal Hospital, Bangalore, Karnataka
  - Srinivasam Cancer Care Multispeciality Hospitals India Pvt Ltd, Bangalore, Karnataka
  - Sahyadri Clinical Research and Development Centre, Pune, Maharashtra
  - Sahyadri Specialty Hospital, Pune, Maharashtra
- Italy (14):
  - AOU Policlinico Vittorio Emanuele-P.O.G. Rodolico, Catania, CT
  - ASST Monza - A.O. San Gerardo, Monza, MB
  - IRCCS Ospedale San Raffaele, Milan, MI
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - Istituto Europeo di Oncologia, Milan, MI
  - Istituto Clinico Humanitas, Rozzano, MI
  - Azienda Ospedaliera di Perugia - Ospedale S. M. Misericordia, Perugia, PG
  - Centro di Riferimento Oncologico-IRCCS, Pordenone, PN
  - Azienda Ospedaliero-Universitaria di Parma, Parma, PR
  - Istituto Nazionale Tumori Regina Elena, Roma, RM
  - Az.Osp.San Camillo-Forlanini, Roma, RM
  - Azienda Ospedaliera Dei Colli Ospedale Monaldi, Napoli
  - Istituto Nazionale Tumori di Napoli, Napoli
  - Ausl della Romagna- Ravenna, Ravenna
- Japan (19):
  - Aichi cancer center central hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
  - National Hospital Organization, Yamaguchi-Ube Medical Center, Ube, Yamaguchi
  - The Cancer Institute Hospital of JFCR, Kōtoku
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - Tokushima University Hospital, Tokushima
  - Wakayama Medical University Department of Pulmonary Medicine and Oncology, Wakayama
- Mexico (3):
  - Médicos Especialistas en Cancer S.C. / San Peregrino., Aguascalientes
  - Instituto Nacional de Cancerologia, Distrito Federal
  - Instituto Nacional de Enfermedades Respiratorias Ismael Cosio Villegas, Distrito Federal
- University Medical Center Groningen, Groningen, Netherlands
- Poland (4):
  - Klinika Onkologii i Radioterapii Uniwersyteckie Centrum Kliniczne, Gdansk
  - Med-Polonia Sp. z o.o., Poznan
  - Centrum Medyczne Dom Lekarski S.A., Szczecin
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie-Panstwowy Instytut Badawczy, Warsaw
- Russia (6):
  - RBHI Kursk Regional Clinical Oncology Dispensary, Kislino, Kursk Oblast
  - Budgetary Healthcare Institution Omsk Region "Clinical Oncological Dispensary", Omsk, Omsk Oblast
  - LEC at SBIH "Saint-Petersburg Clinical Research Practical Center of specialized types of, Pesochniy Poselok, Sankt-Peterburg
  - Private Medical Institution "Euromedservice", Pushkin, Sankt-Peterburg
  - RBHI Kursk Regional Clinical Oncology Dispensary, Kursk
  - FSBI "N.N.Blokhin Medical Research Center of Oncology", Moscow
- Singapore (2):
  - National University Hospital, Singapore
  - Raffles Hospital, Singapore
- South Korea (5):
  - The Catholic University of Korea, St. Vincents Hospital, Suwon, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Division of Medical Oncology, Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (13):
  - Institut Catala d'Oncologia L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Complejo Hospitalario De Navarra, Pamplona, Navarre
  - Hospital Teresa Herrera C.H.U.A.C., A Coruña
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Institut Catala d'Oncologia Girona, Girona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Fe, Valencia
- Taiwan (5):
  - National Taiwan University Hospital, Taipei, Taiwan ROC
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (4):
  - Cukurova University Medical Faculty, Adana
  - Istanbul University Oncology Institute, Istanbul
  - Marmara Univ Pendik Training and Research Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
- United Kingdom (3):
  - The Ipswich Hospital NHS Trust, Ipswich, Suffolk
  - Heart of England NHS Foundation Trust, Birmingham Heartlands Hospital, Birmingham, WEST Midlands
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Liu G, Solomon BJ, Mazieres J, Kim DW, Cortinovis D, Inoue T, Sharma R, Thurm H, Polli A, Bauer TM. Kinetics and management of adverse events associated with lorlatinib after 5 years of follow-up in the CROWN study. Oncologist. 2025 Oct 1;30(10):oyaf287. doi: 10.1093/oncolo/oyaf287. PMID 41124598
- [Derived] Wu YL, Kim HR, Soo RA, Zhou Q, Akamatsu H, Chang GC, Chiu CH, Hayashi H, Kim SW, Goto Y, Kato T, Zhou J, Lee VH, Nishio M, Han B, Kim DW, Lu S, Polli A, Martini JF, Toffalorio F, Wong CH, Mok T. First-Line Lorlatinib Versus Crizotinib in Asian Patients With Advanced ALK-Positive NSCLC: Five-Year Outcomes From the CROWN Study. J Thorac Oncol. 2025 Jul;20(7):955-968. doi: 10.1016/j.jtho.2025.02.021. Epub 2025 Feb 28. PMID 40024442
- [Derived] Solomon BJ, Liu G, Felip E, K Mok TS, Soo RA, Mazieres J, Shaw AT, Marinis F, Goto Y, Wu YL, Kim DW, Martini JF, Messina R, Paolini J, Polli A, Thomaidou D, Toffalorio F, Bauer TM. Plain language summary: 5-year results from the CROWN study of lorlatinib vs crizotinib in non-small-cell lung cancer. Future Oncol. 2024 Dec;20(40):3377-3387. doi: 10.1080/14796694.2024.2406117. Epub 2024 Oct 3. PMID 39360949
- [Derived] Solomon BJ, Liu G, Felip E, Mok TSK, Soo RA, Mazieres J, Shaw AT, de Marinis F, Goto Y, Wu YL, Kim DW, Martini JF, Messina R, Paolini J, Polli A, Thomaidou D, Toffalorio F, Bauer TM. Lorlatinib Versus Crizotinib in Patients With Advanced ALK-Positive Non-Small Cell Lung Cancer: 5-Year Outcomes From the Phase III CROWN Study. J Clin Oncol. 2024 Oct 10;42(29):3400-3409. doi: 10.1200/JCO.24.00581. Epub 2024 May 31. PMID 38819031
- [Derived] Soo RA, Martini JF, van der Wekken AJ, Teraoka S, Ferrara R, Shaw AT, Shepard D, Calella AM, Polli A, Toffalorio F, Tomasini P, Chiu CH, Kowalski DM, Kim HR, Solomon BJ. Early Circulating Tumor DNA Dynamics and Efficacy of Lorlatinib in Patients With Treatment-Naive, Advanced, ALK-Positive NSCLC. J Thorac Oncol. 2023 Nov;18(11):1568-1580. doi: 10.1016/j.jtho.2023.05.021. Epub 2023 Jun 7. PMID 37295609
- [Derived] Solomon BJ, Bauer TM, Mok TSK, Liu G, Mazieres J, de Marinis F, Goto Y, Kim DW, Wu YL, Jassem J, Lopez FL, Soo RA, Shaw AT, Polli A, Messina R, Iadeluca L, Toffalorio F, Felip E. Efficacy and safety of first-line lorlatinib versus crizotinib in patients with advanced, ALK-positive non-small-cell lung cancer: updated analysis of data from the phase 3, randomised, open-label CROWN study. Lancet Respir Med. 2023 Apr;11(4):354-366. doi: 10.1016/S2213-2600(22)00437-4. Epub 2022 Dec 16. PMID 36535300
- [Derived] Solomon BJ, Bauer TM, Ignatius Ou SH, Liu G, Hayashi H, Bearz A, Penkov K, Wu YL, Arrieta O, Jassem J, Calella AM, Peltz G, Polli A, Thurm H, Mok T. Post Hoc Analysis of Lorlatinib Intracranial Efficacy and Safety in Patients With ALK-Positive Advanced Non-Small-Cell Lung Cancer From the Phase III CROWN Study. J Clin Oncol. 2022 Nov 1;40(31):3593-3602. doi: 10.1200/JCO.21.02278. Epub 2022 May 23. PMID 35605188
- [Derived] Solomon BJ, Bauer TM, de Marinis F, Felip E, Goto Y, Liu G, Mazieres J, Kim DW, Mok T, Polli A, Thurm H, Calella AM, Peltz G, Shaw AT. Plain language summary of the CROWN study comparing lorlatinib with crizotinib for people with untreated non-small cell lung cancer. Future Oncol. 2021 Dec 1;17(34):4649-4656. doi: 10.2217/fon-2021-0904. Epub 2021 Sep 29. PMID 34585621
- [Derived] Shaw AT, Bauer TM, de Marinis F, Felip E, Goto Y, Liu G, Mazieres J, Kim DW, Mok T, Polli A, Thurm H, Calella AM, Peltz G, Solomon BJ; CROWN Trial Investigators. First-Line Lorlatinib or Crizotinib in Advanced ALK-Positive Lung Cancer. N Engl J Med. 2020 Nov 19;383(21):2018-2029. doi: 10.1056/NEJMoa2027187. PMID 33207094
- [Derived] Shaw AT, Felip E, Bauer TM, Besse B, Navarro A, Postel-Vinay S, Gainor JF, Johnson M, Dietrich J, James LP, Clancy JS, Chen J, Martini JF, Abbattista A, Solomon BJ. Lorlatinib in non-small-cell lung cancer with ALK or ROS1 rearrangement: an international, multicentre, open-label, single-arm first-in-man phase 1 trial. Lancet Oncol. 2017 Dec;18(12):1590-1599. doi: 10.1016/S1470-2045(17)30680-0. Epub 2017 Oct 23. PMID 29074098
- [Derived] Gainor JF, Shaw AT. J-ALEX: alectinib versus crizotinib in ALK-positive lung cancer. Lancet. 2017 Jul 1;390(10089):3-4. doi: 10.1016/S0140-6736(17)31074-7. Epub 2017 May 10. No abstract available. PMID 28501139
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase 3, randomized, open label study was conducted at 104 sites in 23 countries. A total of 296 participants were randomized, 149 to the lorlatinib arm and 147 to the crizotinib arm.
Pre-assignment Details: Previously untreated Stage IIIB/IV participants with ALK-positive non-small cell lung cancer were randomized in this study.
Groups:
- Lorlatinib: Lorlatinib monotherapy at the recommended Phase 2 dose of 100 mg, was administered orally once daily (QD) at approximately the same time of the day on a continuous daily dosing schedule. Each treatment cycle was defined as 28 days. Treatment continued until confirmation of RECIST version 1.1 defined disease progression assessed by the blinded independent central review (unless clinical benefit was still achievable), participant refusal, participant lost to follow-up, unacceptable toxicity, death, or the study was terminated by the sponsor, whichever occurred first.
- Crizotinib: Crizotinib monotherapy at the registered dose of 250 mg, was administered orally twice daily (BID) at approximately the same time in the morning and evening (12 hours apart) on a continuous daily dosing schedule. Each treatment cycle was defined as 28 days. Treatment continued until confirmation of RECIST version 1.1 defined disease progression assessed by the blinded independent central review (unless clinical benefit was still achievable), participant refusal, participant lost to follow-up, unacceptable toxicity, death, or the study was terminated by the sponsor, whichever occurred first.
Period: Treatment Phase
Arm/Group | Lorlatinib | Crizotinib
Started | 149 | 147
Completed ("Completed" refers to participants with confirmed RECIST version 1.1 defined disease progression assessed by the blinded independent central review or investigator.) | 26 | 83
Not Completed | 123 | 64
Not completed — Adverse Event | 10 | 12
Not completed — Death | 6 | 4
Not completed — Withdrawal by Subject | 4 | 12
Not completed — Global Deterioration of Health Status | 0 | 3
Not completed — Subject decided to continue study treatment as per clinical practice in another hospital. | 0 | 1
Not completed — Subject didn't receive study treatment. | 0 | 1
Not completed — Ongoing | 103 | 31
Period: Long-Term Follow-up Phase
Arm/Group | Lorlatinib | Crizotinib
Started (The long-term follow-up phase included the post-treatment follow-up and the survival follow-up. Participants who started the long-term follow-up phase consisted of participants in both the post-treatment follow-up and the survival follow-up.) | 149 | 147
Completed | 0 | 0
Not Completed | 149 | 147
Not completed — Death | 23 | 28
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 4 | 18
Not completed — Ongoing | 122 | 99

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lorlatinib | Crizotinib | Total
Number analyzed (Participants) | 149 | 147 | 296
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.1 (13.12) | 55.6 (13.52) | 57.4 (13.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 91 | 175
  Male | 65 | 56 | 121
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 72 | 72 | 144
  Race: Black or African American | 0 | 1 | 1
  Race: Asian | 65 | 65 | 130
  Race: Missing | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Based on Blinded Independent Central Review (BICR) Assessment
Description: PFS was defined as the time from randomization to the date of the first documentation of progressive disease as assessed by the independent radiologist or death due to any cause, whichever occurred first. PFS (in months) was calculated as (date of event or censoring-randomization+1)/30.4375. Progressive disease is defined per RECIST version 1.1, as at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of 1 or more new lesions.
Time Frame: From time of Study Start up to 33 months
Population: The full analysis (FA) population included all participants who were randomized, and participants were classified according to the treatment assigned at randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 149 | 147
Months | NA [NA to NA] — The values were not estimable because there were insufficient events to estimate the median PFS time and 95% confidence interval. | 9.3 [7.6 to 11.1]
Statistical Analysis 1: Comparison: Lorlatinib vs Crizotinib; The study was designed to test the null hypothesis H0: λ ≥1 versus the alternative hypothesis HA: λ <1, where λ is the hazard ratio (HR; Lorlatinib/Crizotinib). Evaluation of 177 PFS events was required to have at least 90% power to detect a HR of 0.611 using a one-sided stratified log-rank test at a significance level of 0.025 (one-sided), and a 2-look group-sequential design with a Lan-DeMets (O'Brien-Fleming) α-spending function to determine the efficacy boundaries; Test type: Superiority; p < 0.0001, one-sided stratified log-rank — The study was to be considered positive if the 1-sided log-rank test for PFS, stratified for baseline stratification factors (ethnicity and brain metastases) was significant at the 0.0081 level at the cutoff date of this report; Stratified by the presence of brain metastases (Yes/No) and ethnic origin (Asian/Non-Asian) at randomization; Hazard Ratio (HR) = 0.28, 95% CI 2-sided [0.191 to 0.413] — Based on Cox Proportional Hazards model stratified by the presence of brain metastases and ethnic origin at randomization. Assuming proportional hazards, a hazard ratio less than 1 indicates a reduction in hazard rate in favor of Lorlatinib

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death due to any cause. OS (in months) was calculated as (date of death or censoring - start date +1)/30.4375. Participants last known to be alive were censored at date of last contact.
Time Frame: From time of Study Start up to 33 months
Population: The FA population included all participants who were randomized, and participants were classified according to the treatment assigned at randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 149 | 147
Months | NA [NA to NA] — The values were not estimable because there were insufficient events to estimate the median OS time and 95% confidence interval. | NA [NA to NA] — The values were not estimable because there were insufficient events to estimate the median OS time and 95% confidence interval.
Statistical Analysis 1: Comparison: Lorlatinib vs Crizotinib; Test type: Superiority; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.414 to 1.249] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Progression-Free Survival (PFS) Based on Investigator's Assessment
Description: PFS was defined as the time from randomization to the date of the first documentation of progressive disease as assessed by investigator or death due to any cause, whichever occurred first. PFS (in months) was calculated as (date of event or censoring-randomization+1)/30.4375. Progressive disease is defined per RECIST version 1.1, as at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of 1 or more new lesions.
Time Frame: From time of Study Start up to 33 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 149 | 147
Months | NA [NA to NA] — The values were not estimable because there were insufficient events to estimate the median PFS time and 95% confidence interval. | 9.1 [7.4 to 10.9]
Statistical Analysis 1: Comparison: Lorlatinib vs Crizotinib; Test type: Superiority; p < 0.0001, one-sided stratified log-rank; Stratified by the presence of brain metastases (Yes/No) and ethnic origin (Asian/Non-Asian) at randomization; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.144 to 0.307] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Objective Response Rate (ORR) - Percentage of Participants With Objective Response (OR) Based on BICR Assessment
Description: ORR was the percentage of participants with objective response of complete response (CR) or partial response (PR) according to RECIST version 1.1 recorded from randomization until disease progression or start of new anti-cancer therapy. CR was defined as complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). PR was defined as at least a 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: From time of Study Start up to 33 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 149 | 147
Percentage of participants | 75.8 [68.2 to 82.5] | 57.8 [49.4 to 65.9]
Statistical Analysis 1: Comparison: Lorlatinib vs Crizotinib; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel; Stratified by the presence of brain metastases (Yes/No) and ethnic origin (Asian/Non-Asian) at randomization; Odds Ratio (OR) = 2.254, 95% CI 2-sided [1.353 to 3.891] — Odds ratio was estimated using Mantel-Haenszel method. An odds ratio larger than 1 indicates better outcome for Lorlatinib relative to Crizotinib. Exact CI was calculated

5. Secondary Outcome: Objective Response Rate (ORR) - Percentage of Participants With Objective Response (OR) Based on Investigator's Assessment
Description: as for outcome 4
Time Frame: From time of Study Start up to 33 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 149 | 147
Percentage of participants | 80.5 [73.3 to 86.6] | 61.9 [53.5 to 69.8]
Statistical Analysis 1: Comparison: Lorlatinib vs Crizotinib; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Stratified by the presence of brain metastases (Yes/No) and ethnic origin (Asian/Non-Asian) at randomization; Odds Ratio (OR) = 2.499, 95% CI 2-sided [1.484 to 4.594] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Intracranial Objective Response Rate (IC-ORR) - Percentage of Participants With Intracranial Objective Response (IC-OR) Based on BICR Assessment
Description: IC-ORR was the percentage of participant with intracranial objective response of complete response (CR) or partial response (PR) based on intracranial disease in the subset of participants with at least 1 intracranial lesion per RECIST version 1.1 (modified) recorded from randomization until disease progression or start of new anti-cancer therapy. CR was defined as complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). PR was defined as at least a 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: From time of Study Start up to 33 months
Population: The subset of the FA population with at least 1 baseline intracranial lesion (based on BICR intracranial assessment).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 38 | 40
Percentage of participants | 65.8 [48.6 to 80.4] | 20.0 [9.1 to 35.6]
Statistical Analysis 1: Comparison: Lorlatinib vs Crizotinib; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by the presence of brain metastases (Yes/No) and ethnic origin (Asian/Non-Asian) at randomization; Odds Ratio (OR) = 8.407, 95% CI 2-sided [2.586 to 27.233] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Intracranial Time to Progression (IC-TTP) Based on BICR Assessment
Description: IC-TTP based on BICR assessment was defined as the time from date of randomization to the date of the first documentation of progression of intracranial disease, based on either new brain metastases or progression of existing brain metastases.
Time Frame: From time of Study Start up to 33 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 149 | 147
Months | NA [NA to NA] — The values were not estimable because there were insufficient events to estimate the median IC-TTP time and 95% confidence interval. | 16.6 [11.1 to NA] — The value was not estimable because there were insufficient events to estimate the upper bound of the 95% confidence interval.
Statistical Analysis 1: Comparison: Lorlatinib vs Crizotinib; Test type: Superiority; p < 0.0001, one-sided stratified log-rank; Stratified by the presence of brain metastases (Yes/No) and ethnic origin (Asian/Non-Asian) at randomization; Hazard Ratio (HR) = 0.07, 95% CI 2-sided [0.026 to 0.170] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Duration of Response (DR) Based on BICR Assessment
Description: DR was defined, for participants with a confirmed objective response (OR) of complete response (CR) or partial response (PR) per RECIST version 1.1, as the time from the first documentation of OR to the first documentation of progressive disease (PD) or death due to any cause, whichever occurred first. CR was defined as complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). PR was defined as at least a 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. PD was defined as at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of 1 or more new lesions.
Time Frame: From time of Study Start up to 33 months
Population: Participants with a confirmed objective response (complete response or partial response) per RECIST version 1.1 in the FA population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 113 | 85
Months | NA [NA to NA] — The values were not estimable because there were insufficient events to estimate the median DR time and the 95% confidence interval. | 11.0 [9.0 to 12.9]

9. Secondary Outcome: Intracranial Duration of Response (IC-DR) Based on BICR Assessment
Description: IC-DR was defined, for participants with a confirmed intracranial objective response (OR) of complete response (CR) or partial response (PR) per RECIST version 1.1, as the time from the first documentation of intracranial OR to the first documentation of intracranial progressive disease (PD) or death due to any cause, whichever occurred first. CR was defined as complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). PR was defined as at least a 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. PD was defined as at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of 1 or more new lesions.
Time Frame: From time of Study Start up to 33 months
Population: Participants with brain metastases at baseline and confirmed intracranial complete response or partial response in the FA population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 25 | 8
Months | NA [NA to NA] — The values were not estimable because there were insufficient events to estimate the median IC-DR time and the 95% confidence interval. | 9.4 [6.0 to 11.1]

10. Secondary Outcome: Time to Tumor Response (TTR) Based on BICR Assessment
Description: TTR based on BICR assessment was defined, for participants with a confirmed objective response, as the time from the date of randomization to the first documentation of objective response (complete response or partial response) which was subsequently confirmed. Complete response was defined as complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). Partial response was defined as at least a 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: From time of Study Start up to 33 months
Population: Participants with confirmed complete response or partial response in the FA population.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 113 | 85
Months | 1.8 [1.7 to 1.9] | 1.8 [1.7 to 1.9]

11. Secondary Outcome: Intracranial Time to Tumor Response (IC-TTR) Based on BICR Assessment
Description: IC-TTR was defined, for participants with a confirmed intracranial objective response, as the time from the date of randomization to the first documentation of intracranial objective response (complete response or partial response) which was subsequently confirmed. Complete response was defined as complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). Partial response was defined as at least a 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: From time of Study Start up to 33 months
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 25 | 8
Months | 1.9 [1.8 to 3.7] | 1.8 [1.7 to 2.7]

12. Secondary Outcome: PFS2 Based on Investigator's Assessment
Description: PFS2 was defined as the time from randomization to the date of progression of disease on first subsequent systemic anti-cancer therapy, or death from any cause, whichever occurred first
Time Frame: From time of Study Start up to 45 months
Reporting Status: Not Posted, anticipated posting 2027-12

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs; All-Causality and Treatment-Related)
Description: An AE was an untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes: death, life-threatening experience, initial or prolonged inpatient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect. Treatment-emergent AEs were those with initial onset or that worsen in severity after the first dose of study medication. All AEs in the table below were treatment-emergent AEs. Grade 3 and 4 AEs in the table below indicated severe AE and life-threatening consequences respectively; Grade 5 indicated death due to AE. Treatment-related AEs were determined by investigators.
Time Frame: From time of Study Start up to 33 months
Population: The safety analysis population included all participants who received at least 1 dose of study drug. Participants were classified according to the treatment assigned at randomization unless the incorrect treatment(s) were received throughout the dosing period, in which case participants were classified according to the first study treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 149 | 142
Participants
  AEs (all-causality) | 149 | 140
  AEs (treatment-related) | 144 | 133
  SAEs (all-causality) | 51 | 39
  SAEs (treatment-related) | 12 | 7
  Maximum Grade 3 or 4 AEs (all-causality) | 108 | 79
  Maximum Grade 3 or 4 AEs (treatment-related) | 83 | 52
  Maximum Grade 5 AEs (all-causality) | 7 | 7
  Maximum Grade 5 AEs (treatment-related) | 2 | 0
  AEs causing study discontinuation (all-causality) | 7 | 8
  AEs causing study discontinuation (treatment-related) | 2 | 0
  AEs causing study treatment discontinuation (all-causality) | 10 | 13
  AEs causing study treatment discontinuation (treatment-related) | 7 | 7
  AEs causing dose reduction or temporary discontinuation (all-causality) | 79 | 71
  AEs causing dose reduction or temporary discontinuation (treatment-related) | 60 | 54

14. Secondary Outcome: Number of Participants With Changes in Hematology Laboratory Parameters From Baseline Maximum NCI-CTCAE Grade Lower Than 3 to Postbaseline Maximum Grade 3 or Grade 4
Description: Laboratory test results were graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grades 1 and 2 indicate mild and moderate AE, respectively; Grades 3 and 4 indicate severe AE and life-threatening consequences respectively; Grade 5 indicates death due to AE. Participants with laboratory test abnormalities were summarized according to the worst grade for each laboratory test result. All participants meeting the postbaseline grade criteria in the table below had baseline maximum grades lower than 3.
Time Frame: From Baseline up to 33 months
Population: Participants in the safety analysis population who had at least one on-study assessment for the parameter of interest.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 149 | 141
Participants
  Anemia (Postbaseline Maximum Grade 3) | 3 | 4
  Anemia (Postbaseline Maximum Grade 4) | NA — CTCAE grade not defined. | NA — CTCAE grade not defined.
  Hemoglobin increased (Postbaseline Maximum Grade 3) | 0 | 0
  Hemoglobin increased (Postbaseline Maximum Grade 4) | NA — CTCAE grade not defined. | NA — CTCAE grade not defined.
  Lymphocyte count decreased (Postbaseline Maximum Grade 3) | 2 | 7
  Lymphocyte count decreased (Postbaseline Maximum Grade 4) | 2 | 1
  Lymphocyte count increased (Postbaseline Maximum Grade 3) | 0 | 0
  Lymphocyte count increased (Postbaseline Maximum Grade 4) | NA — CTCAE grade not defined. | NA — CTCAE grade not defined.
  Neutrophil count decreased (Postbaseline Maximum Grade 3) | 1 | 19
  Neutrophil count decreased (Postbaseline Maximum Grade 4) | 1 | 4
  Platelet count decreased (Postbaseline Maximum Grade 3) | 0 | 1
  Platelet count decreased (Postbaseline Maximum Grade 4) | 0 | 0
  White blood cell decreased (Postbaseline Maximum Grade 3) | 0 | 5
  White blood cell decreased (Postbaseline Maximum Grade 4) | 0 | 0

15. Secondary Outcome: Number of Participants With Changes in Chemistry Laboratory Parameters From Baseline Maximum NCI-CTCAE Grade Lower Than 3 to Postbaseline Maximum Grade 3 or Grade 4
Description: as for outcome 14
Time Frame: From Baseline up to 33 months
Population: Participants in the safety analysis population who had at least one on-study assessment for the parameter of interest.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 149 | 141
Participants
  Alanine aminotransferase increased (Postbaseline Maximum Grade 3) | 4 | 5
  Alanine aminotransferase increased (Postbaseline Maximum Grade 4) | 0 | 1
  Alkaline phosphate increased (Postbaseline Maximum Grade 3) | 0 | 1
  Alkaline phosphate increased (Postbaseline Maximum Grade 4) | 0 | 0
  Aspartate aminotransferase increased (Postbaseline Maximum Grade 3) | 3 | 4
  Aspartate aminotransferase increased (Postbaseline Maximum Grade 4) | 0 | 1
  Blood bilirubin increased (Postbaseline Maximum Grade 3) | 0 | 0
  Blood bilirubin increased (Postbaseline Maximum Grade 4) | 0 | 0
  Creatine kinase increased (Postbaseline Maximum Grade 3) | 3 | 5
  Creatine kinase increased (Postbaseline Maximum Grade 4) | 0 | 2
  Creatinine increased (Postbaseline Maximum Grade 3) | 1 | 3
  Creatinine increased (Postbaseline Maximum Grade 4) | 0 | 0
  Gamma glutamyl transferase increased (Postbaseline Maximum Grade 3) | 9 | 8
  Gamma glutamyl transferase increased (Postbaseline Maximum Grade 4) | 0 | 1
  Hypercalcemia (Postbaseline Maximum Grade 3) | 0 | 0
  Hypercalcemia (Postbaseline Maximum Grade 4) | 0 | 0
  Hyperglycemia (Postbaseline Maximum Grade 3) | 9 | 3
  Hyperglycemia (Postbaseline Maximum Grade 4) | 1 | 0
  Hyperkalemia (Postbaseline Maximum Grade 3) | 2 | 3
  Hyperkalemia (Postbaseline Maximum Grade 4) | 0 | 0
  Hypermagnesemia (Postbaseline Maximum Grade 3) | 2 | 1
  Hypermagnesemia (Postbaseline Maximum Grade 4) | 0 | 0
  Hypernatremia (Postbaseline Maximum Grade 3) | 0 | 0
  Hypernatremia (Postbaseline Maximum Grade 4) | 0 | 0
  Hypoalbuminemia (Postbaseline Maximum Grade 3) | 1 | 9
  Hypoalbuminemia (Postbaseline Maximum Grade 4) | NA — CTCAE grade not defined. | NA — CTCAE grade not defined.
  Hypocalcemia (Postbaseline Maximum Grade 3) | 1 | 0
  Hypocalcemia (Postbaseline Maximum Grade 4) | 0 | 0
  Hypoglycemia (Postbaseline Maximum Grade 3) | 0 | 0
  Hypoglycemia (Postbaseline Maximum Grade 4) | 0 | 1
  Hypokalemia (Postbaseline Maximum Grade 3) | 0 | 3
  Hypokalemia (Postbaseline Maximum Grade 4) | 0 | 0
  Hypomagnesemia (Postbaseline Maximum Grade 3) | 0 | 0
  Hypomagnesemia (Postbaseline Maximum Grade 4) | 0 | 0
  Hyponatremia (Postbaseline Maximum Grade 3) | 5 | 10
  Hyponatremia (Postbaseline Maximum Grade 4) | 0 | 1
  Hypophosphatemia (Postbaseline Maximum Grade 3) | 3 | 4
  Hypophosphatemia (Postbaseline Maximum Grade 4) | 0 | 0
  Lipase increased (Postbaseline Maximum Grade 3) | 8 | 6
  Lipase increased (Postbaseline Maximum Grade 4) | 3 | 1
  Serum amylase increased (Postbaseline Maximum Grade 3) | 1 | 2
  Serum amylase increased (Postbaseline Maximum Grade 4) | 0 | 0

16. Secondary Outcome: Number of Participants With Changes in Lipid Laboratory Parameters From Baseline Maximum NCI-CTCAE Grade Lower Than 3 to Postbaseline Maximum Grade 3 or Grade 4
Description: as for outcome 14
Time Frame: From Baseline up to 33 months
Population: Participants in the safety analysis population who had at least one on-study assessment for the parameter of interest.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 149 | 141
Participants
  Cholesterol high (Postbaseline Maximum Grade 3) | 26 | 0
  Cholesterol high (Postbaseline Maximum Grade 4) | 3 | 0
  Hypertriglyceridemia (Postbaseline Maximum Grade 3) | 20 | 0
  Hypertriglyceridemia (Postbaseline Maximum Grade 4) | 13 | 0

17. Secondary Outcome: Number of Participant With Vital Signs and Body Weight Data Meeting Pre-defined Criteria
Description: Vital signs data included pulse, systolic blood pressure, and diastolic blood pressure. Measurements were only provided once per timepoint. If multiple assessments were provided per timepoint, the maximum value were used for reporting. The pre-defined criteria of vital sign and body weight data were as follows: maximum pulse rate >120 beats per minute (bpm); minimum pulse rate <50 bpm; maximum increase in pulse rate ≥30 bpm; maximum decrease in pulse rate ≥30 bpm; increase in systolic blood Pressure ≥40 mmHg; decrease in systolic blood pressure ≥40 mmHg; decrease in systolic blood pressure ≥60 mmHg; increase in diastolic blood pressure ≥20 mmHg; decrease in diastolic blood pressure ≥20 mmHg; decrease in diastolic blood pressure ≥40 mmHg; increase in body weight ≥10%; increase in body weight ≥20%; decrease in body weight ≥10%.
Time Frame: From Baseline up to 33 months
Population: "Number of Participants Analyzed" included all participants in the safety analysis population. "Number Analyzed" included all participants in the safety analysis population with evaluable data against the pre-defined criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 149 | 142
Participants
  Sitting pulse rate: pulse >120 bpm | 7 | 1
  Sitting pulse rate: pulse <50 bpm | 4 | 22
  Sitting pulse rate: change ≥30 bpm increase: number analyzed (Participants) | 147 | 142
  Sitting pulse rate: change ≥30 bpm increase | 24 | 3
  Sitting pulse rate: change ≥30 bpm decrease: number analyzed (Participants) | 147 | 142
  Sitting pulse rate: change ≥30 bpm decrease | 17 | 47
  Sitting systolic blood pressure: change ≥40 mmHg increase: number analyzed (Participants) | 147 | 142
  Sitting systolic blood pressure: change ≥40 mmHg increase | 22 | 3
  Sitting systolic blood pressure: change ≥40 mmHg decrease: number analyzed (Participants) | 147 | 142
  Sitting systolic blood pressure: change ≥40 mmHg decrease | 6 | 14
  Sitting systolic blood pressure: change ≥60 mmHg decrease: number analyzed (Participants) | 147 | 142
  Sitting systolic blood pressure: change ≥60 mmHg decrease | 0 | 1
  Sitting diastolic blood pressure: change ≥20 mmHg increase: number analyzed (Participants) | 147 | 142
  Sitting diastolic blood pressure: change ≥20 mmHg increase | 41 | 18
  Sitting diastolic blood pressure: change ≥20 mmHg decrease: number analyzed (Participants) | 147 | 142
  Sitting diastolic blood pressure: change ≥20 mmHg decrease | 26 | 52
  Sitting diastolic blood pressure: change ≥40 mmHg decrease: number analyzed (Participants) | 147 | 142
  Sitting diastolic blood pressure: change ≥40 mmHg decrease | 0 | 1
  Body weight (kg): percent change from baseline ≥10% increase: number analyzed (Participants) | 146 | 137
  Body weight (kg): percent change from baseline ≥10% increase | 99 | 39
  Body weight (kg): percent change from baseline ≥20% increase: number analyzed (Participants) | 146 | 137
  Body weight (kg): percent change from baseline ≥20% increase | 35 | 3
  Body weight (kg): percent change from baseline ≥10% decrease: number analyzed (Participants) | 146 | 137
  Body weight (kg): percent change from baseline ≥10% decrease | 6 | 12

18. Secondary Outcome: Number of Participant With Maximum Increase From Baseline in Electrocardiogram (ECG) Data Meeting Pre-defined Criteria
Description: Baseline was defined as the last assessment performed on or prior to date of the first dose of study treatment. Triplicate ECGs were collected in the study and the average of the replicate assessments were used for summary analysis. The pre-defined criteria of ECG data were as follows: change from baseline in QTcF ≥60 msec, ≥30 msec but <60 msec, <30 msec; change from baseline in QTcB ≥60 msec, ≥30 msec but <60 msec, <30 msec; PR change ≥50% if absolute baseline value was <200 msec; PR change ≥25% if absolute baseline value was ≥200 msec; QRS change ≥50% if absolute baseline value was <100 msec; QRS change ≥25% if absolute baseline value was ≥100 msec.
Time Frame: From Baseline up to 33 months
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 149 | 142
Participants
  Change of QTcF ≥60 msec: number analyzed (Participants) | 146 | 138
  Change of QTcF ≥60 msec | 5 | 16
  30 msec ≤ Change of QTcF <60 msec: number analyzed (Participants) | 146 | 138
  30 msec ≤ Change of QTcF <60 msec | 49 | 41
  Change of QTcF <30 msec: number analyzed (Participants) | 146 | 138
  Change of QTcF <30 msec | 92 | 81
  Change of QTcB ≥60 msec: number analyzed (Participants) | 149 | 141
  Change of QTcB ≥60 msec | 10 | 15
  30 msec ≤ Change of QTcB <60 msec: number analyzed (Participants) | 149 | 141
  30 msec ≤ Change of QTcB <60 msec | 49 | 26
  Change of QTcB <30 msec: number analyzed (Participants) | 149 | 141
  Change of QTcB <30 msec | 90 | 100
  PR change ≥50% if absolute baseline value was <200 msec: number analyzed (Participants) | 146 | 140
  PR change ≥50% if absolute baseline value was <200 msec | 8 | 4
  PR change ≥25% if absolute baseline value was ≥200 msec: number analyzed (Participants) | 146 | 140
  PR change ≥25% if absolute baseline value was ≥200 msec | 0 | 0
  QRS change ≥50% if absolute baseline value was <100 msec: number analyzed (Participants) | 149 | 141
  QRS change ≥50% if absolute baseline value was <100 msec | 2 | 3
  QRS change ≥25% if absolute baseline value was ≥100 msec: number analyzed (Participants) | 149 | 141
  QRS change ≥25% if absolute baseline value was ≥100 msec | 2 | 0

19. Secondary Outcome: Number of Participants With Maximum Decrease From Baseline Greater Than or Equal to 20 Points in Left Ventricular Ejection Fraction (LVEF) Percentage
Description: In this outcome measure, baseline was defined as the last assessment on or prior to the date of the first dose of study treatment. Decrease from baseline was an absolute difference between baseline and observed value.
Time Frame: From Baseline up to 33 months
Population: All participants in the safety analysis population who had at least one on-study assessment for the parameter of interest.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 143 | 133
Participants | 2 | 1

20. Secondary Outcome: Change From Baseline in Total Scores of Beck Depression Inventory (BDI)-II (Mood Assessment) Across Time
Description: BDI-II (Mood Assessment) is a 21 item self-reported scale, with each item rated by participants on a 4-point scale (ranging from 0-3). The scale includes items capturing mood, (loss of pleasure, sadness, and irritability), suicidal ideation, and cognitive signs (punitive thoughts, self-criticism, self-dislike pessimism, poor concentration) as well as somatic signs (appetite, sleep, fatigue, libido). Scores were obtained by adding up the total points from the series of answers. The total score ranged from 0 to 63, with higher total scores indicating more severe depressive symptoms. The standardized cutoffs are as follows: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; 29-63: severe depression.
Time Frame: Baseline, Cycle 2 Day 1 (C2D1), C3D1, C4D1, C5D1, C6D1, C8D1, C10D1, C12D1, C14D1, C16D1, C18D1, C20D1, C22D1, C24D1, C26D1, C28D1, C30D1, C32D1, C34D1, C36D1, C38D1 and End of Treatment
Population: "Number of Participants Analyzed" included all participants in the safety analysis population within each treatment group. "Number Analyzed" included all participants with at least a baseline and postbaseline assessment at the visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 149 | 147
Units on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 139 | 120
  Cycle 2 Day 1 | -1.8 (5.52) | -1.2 (5.62)
  Cycle 3 Day 1: number analyzed (Participants) | 135 | 115
  Cycle 3 Day 1 | -2.5 (5.85) | -2.7 (5.78)
  Cycle 4 Day 1: number analyzed (Participants) | 127 | 110
  Cycle 4 Day 1 | -2.9 (5.73) | -3.6 (6.60)
  Cycle 5 Day 1: number analyzed (Participants) | 126 | 106
  Cycle 5 Day 1 | -2.5 (6.28) | -3.0 (6.24)
  Cycle 6 Day 1: number analyzed (Participants) | 123 | 96
  Cycle 6 Day 1 | -2.6 (6.61) | -2.9 (6.65)
  Cycle 8 Day 1: number analyzed (Participants) | 123 | 87
  Cycle 8 Day 1 | -3.2 (6.18) | -1.9 (6.56)
  Cycle 10 Day 1: number analyzed (Participants) | 115 | 72
  Cycle 10 Day 1 | -3.0 (6.30) | -2.6 (5.98)
  Cycle 12 Day 1: number analyzed (Participants) | 113 | 58
  Cycle 12 Day 1 | -3.6 (6.05) | -2.1 (6.23)
  Cycle 14 Day 1: number analyzed (Participants) | 108 | 47
  Cycle 14 Day 1 | -3.3 (6.82) | -2.5 (5.57)
  Cycle 16 Day 1: number analyzed (Participants) | 102 | 39
  Cycle 16 Day 1 | -3.3 (6.87) | -2.3 (5.77)
  Cycle 18 Day 1: number analyzed (Participants) | 83 | 28
  Cycle 18 Day 1 | -3.7 (7.26) | -2.6 (4.30)
  Cycle 20 Day 1: number analyzed (Participants) | 67 | 17
  Cycle 20 Day 1 | -3.3 (6.24) | -2.4 (4.62)
  Cycle 22 Day 1: number analyzed (Participants) | 54 | 13
  Cycle 22 Day 1 | -3.2 (6.95) | -2.5 (4.82)
  Cycle 24 Day 1: number analyzed (Participants) | 41 | 9
  Cycle 24 Day 1 | -3.1 (5.97) | 2.3 (9.31)
  Cycle 26 Day 1: number analyzed (Participants) | 33 | 8
  Cycle 26 Day 1 | -3.2 (6.87) | -0.8 (3.81)
  Cycle 28 Day 1: number analyzed (Participants) | 21 | 6
  Cycle 28 Day 1 | -3.0 (6.53) | 0.2 (7.65)
  Cycle 30 Day 1: number analyzed (Participants) | 12 | 4
  Cycle 30 Day 1 | -4.8 (8.00) | 1.3 (3.20)
  Cycle 32 Day 1: number analyzed (Participants) | 8 | 2
  Cycle 32 Day 1 | -5.0 (14.14) | 7.5 (9.19)
  Cycle 34 Day 1: number analyzed (Participants) | 4 | 1
  Cycle 34 Day 1 | -2.3 (12.42) | 0.0
  Cycle 36 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 36 Day 1 |  | 0.0
  Cycle 38 Day 1: number analyzed (Participants) | 0 | 0
  End of Treatment: number analyzed (Participants) | 20 | 60
  End of Treatment | 0.8 (4.49) | -0.2 (7.45)

21. Secondary Outcome: Number of Participants With Suicidal Ideation and Suicidal Behavior Across Time
Description: Suicidal ideation and behaviors were assessed by the Columbia Suicide Severity Rating Scale (C-SSRS). The C-SSRS is a unique, simple and short method of assessing both behavior and ideation that tracks all suicidal events and provides a summary of suicidality. It assesses the lethality of attempts and other features of ideation (frequency, duration, controllability, reasons for ideation, and deterrents), all of which are significantly predictive of completed suicide.
Time Frame: as for outcome 20
Population: "Number of Participants Analyzed" included all participants in the safety analysis population within each treatment group. "Number Analyzed" included all participants with assessment scores at each specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 149 | 142
Participants
  Baseline: number analyzed (Participants) | 147 | 121
  Baseline | 3 | 7
  Cycle 2 Day 1: number analyzed (Participants) | 138 | 119
  Cycle 2 Day 1 | 0 | 5
  Cycle 3 Day 1: number analyzed (Participants) | 137 | 113
  Cycle 3 Day 1 | 1 | 1
  Cycle 4 Day 1: number analyzed (Participants) | 131 | 109
  Cycle 4 Day 1 | 0 | 1
  Cycle 5 Day 1: number analyzed (Participants) | 128 | 103
  Cycle 5 Day 1 | 0 | 1
  Cycle 6 Day 1: number analyzed (Participants) | 123 | 93
  Cycle 6 Day 1 | 0 | 2
  Cycle 8 Day 1: number analyzed (Participants) | 122 | 85
  Cycle 8 Day 1 | 0 | 2
  Cycle 10 Day 1: number analyzed (Participants) | 115 | 68
  Cycle 10 Day 1 | 0 | 1
  Cycle 12 Day 1: number analyzed (Participants) | 114 | 55
  Cycle 12 Day 1 | 0 | 0
  Cycle 14 Day 1: number analyzed (Participants) | 109 | 44
  Cycle 14 Day 1 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 103 | 35
  Cycle 16 Day 1 | 0 | 0
  Cycle 18 Day 1: number analyzed (Participants) | 81 | 25
  Cycle 18 Day 1 | 0 | 0
  Cycle 20 Day 1: number analyzed (Participants) | 67 | 15
  Cycle 20 Day 1 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 54 | 13
  Cycle 22 Day 1 | 0 | 0
  Cycle 24 Day 1: number analyzed (Participants) | 41 | 9
  Cycle 24 Day 1 | 0 | 1
  Cycle 26 Day 1: number analyzed (Participants) | 33 | 8
  Cycle 26 Day 1 | 1 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 23 | 6
  Cycle 28 Day 1 | 0 | 0
  Cycle 30 Day 1: number analyzed (Participants) | 14 | 4
  Cycle 30 Day 1 | 0 | 0
  Cycle 32 Day 1: number analyzed (Participants) | 10 | 2
  Cycle 32 Day 1 | 0 | 0
  Cycle 34 Day 1: number analyzed (Participants) | 6 | 1
  Cycle 34 Day 1 | 0 | 0
  Cycle 36 Day 1: number analyzed (Participants) | 2 | 1
  Cycle 36 Day 1 | 0 | 0
  Cycle 38 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 38 Day 1 | 0 |
  End of Treatment: number analyzed (Participants) | 20 | 62
  End of Treatment | 0 | 0

22. Secondary Outcome: Change From Baseline in Global Quality of Life (QOL), Functional Scales and Symptoms Scales as Assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30) During Overall Treatment
Description: The EORTC QLQ C30 consists of 30 questions and includes 5 functional scales (physical, role, cognitive, emotional, and social); a global health status/global quality of life scale; 3 symptom scales (fatigue, pain, nausea and vomiting); and 6 single items that assess additional symptoms (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea) and financial impact. All scales and single item measures range in score from 0 to 100. Higher scores on the functional scales represent higher levels of functioning. Higher scores on the global health status/quality of life scale represent higher health status/quality of life. Higher scores on symptom scales/items represent a greater presence of symptoms.
Time Frame: From Baseline up to Cycle 38 Day 1
Population: Participants from the FA population who completed a baseline (last patient-reported outcome (PRO) assessment prior to the first dose of study treatment) and at least 1 post-baseline PRO assessment.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 148 | 140
Units on a scale
  Global QOL | 8.60 [6.09 to 11.11] | 3.95 [1.15 to 6.76]
  Physical Functioning | 4.84 [2.67 to 7.01] | 2.82 [0.42 to 5.22]
  Role Functioning | 6.86 [4.05 to 9.68] | 4.78 [1.61 to 7.95]
  Emotional Functioning | 8.77 [6.88 to 10.67] | 6.20 [4.09 to 8.30]
  Cognitive Functioning | -4.20 [-6.56 to -1.84] | -1.02 [-3.64 to 1.60]
  Social Functioning | 7.00 [4.48 to 9.52] | 4.72 [1.87 to 7.57]
  Fatigue | -9.93 [-12.61 to -7.26] | -4.26 [-7.28 to -1.25]
  Nausea and Vomiting | -4.35 [-5.79 to -2.90] | 3.51 [1.89 to 5.14]
  Pain | -4.60 [-7.17 to -2.02] | -5.76 [-8.67 to -2.85]
  Dyspnoea | -7.02 [-9.66 to -4.39] | -8.75 [-11.76 to -5.74]
  Insomnia | -17.34 [-19.71 to -14.96] | -9.39 [-12.07 to -6.71]
  Appetite Loss | -13.15 [-15.00 to -11.30] | -3.95 [-6.01 to -1.88]
  Constipation | -2.40 [-5.33 to 0.54] | 2.53 [-0.83 to 5.90]
  Diarrhea | -0.92 [-3.42 to 1.59] | 11.12 [8.33 to 13.91]
  Financial Difficulties | -6.79 [-9.52 to -4.05] | -5.74 [-8.80 to -2.68]
Statistical Analysis 1: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Global QOL. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.0096, Mixed Models Analysis; Mean Difference (Net) = 4.65, 95% CI 2-sided [1.14 to 8.16]
Statistical Analysis 2: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Physical Functioning. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.1897, Mixed Models Analysis; Mean Difference (Net) = 2.02, 95% CI 2-sided [-1.01 to 5.05]
Statistical Analysis 3: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Role Functioning. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.2999, Mixed Models Analysis; Mean Difference (Net) = 2.09, 95% CI 2-sided [-1.87 to 6.04]
Statistical Analysis 4: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Emotional Functioning. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.0553, Mixed Models Analysis; Mean Difference (Net) = 2.58, 95% CI 2-sided [-0.06 to 5.22]
Statistical Analysis 5: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Cognitive Functioning. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.0588, Mixed Models Analysis; Mean Difference (Net) = -3.18, 95% CI 2-sided [-6.47 to 0.12]
Statistical Analysis 6: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Social Functioning. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.2118, Mixed Models Analysis; Mean Difference (Net) = 2.27, 95% CI 2-sided [-1.30 to 5.85]
Statistical Analysis 7: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Fatigue. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.0032, Mixed Models Analysis; Mean Difference (Net) = -5.67, 95% CI 2-sided [-9.42 to -1.92]
Statistical Analysis 8: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Nausea and Vomiting. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -7.86, 95% CI 2-sided [-9.86 to -5.86]
Statistical Analysis 9: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Pain. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.5310, Mixed Models Analysis; Mean Difference (Net) = 1.16, 95% CI 2-sided [-2.49 to 4.82]
Statistical Analysis 10: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Dyspnoea. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.3602, Mixed Models Analysis; Mean Difference (Net) = 1.72, 95% CI 2-sided [-1.98 to 5.43]
Statistical Analysis 11: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Insomnia. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -7.95, 95% CI 2-sided [-11.25 to -4.64]
Statistical Analysis 12: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Appetite Loss. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -9.21, 95% CI 2-sided [-11.80 to -6.62]
Statistical Analysis 13: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Constipation. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.0198, Mixed Models Analysis; Mean Difference (Net) = -4.93, 95% CI 2-sided [-9.07 to -0.79]
Statistical Analysis 14: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Diarrhea. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -12.03, 95% CI 2-sided [-15.49 to -8.58]
Statistical Analysis 15: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-C30 Financial Difficulties. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.5947, Mixed Models Analysis; Mean Difference (Net) = -1.04, 95% CI 2-sided [-4.90 to 2.82]

23. Secondary Outcome: Change From Baseline in Lung Cancer Symptoms as Assessed by the EORTC Quality of Life Questionnaire-Lung Cancer 13 (QLQ- LC13) During Overall Treatment
Description: The EORTC QLQ LC13 consists of 13 questions and includes 1 multi-item scale and 9 single items assessing symptoms (dyspnea, cough, haemoptysis, and site-specific pain), side effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia), and pain medication use. The scale scores rang from 0 to 100, with higher scores indicating higher ("worse") level of symptoms.
Time Frame: From Baseline up to Cycle 38 Day 1
Population: as for outcome 22
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 146 | 139
Units on a scale
  Dyspnoea | -4.36 [-6.55 to -2.17] | -4.90 [-7.34 to -2.47]
  Coughing | -21.21 [-23.71 to -18.70] | -16.66 [-19.48 to -13.84]
  Haemoptysis | -2.53 [-3.12 to -1.94] | -2.65 [-3.34 to -1.97]
  Sore Mouth | 0.56 [-0.98 to 2.10] | -0.60 [-2.39 to 1.19]
  Dysphagia | -1.35 [-2.95 to 0.25] | 0.16 [-1.68 to 2.00]
  Peripheral Neuropathy | 11.56 [8.21 to 14.91] | 6.20 [2.39 to 10.00]
  Alopecia | 1.61 [-0.97 to 4.20] | 1.81 [-1.08 to 4.70]
  Pain in Chest | -9.54 [-11.27 to -7.80] | -9.01 [-10.97 to -7.05]
  Pain in Arm or Shoulder | -6.93 [-9.43 to -4.43] | -7.38 [-10.24 to -4.52]
  Pain in Other Parts | -2.31 [-5.28 to 0.66] | -5.67 [-8.97 to -2.38]
Statistical Analysis 1: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-LC13 Dyspnoea. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.7254, Mixed Models Analysis; Mean Difference (Net) = 0.55, 95% CI 2-sided [-2.51 to 3.60]
Statistical Analysis 2: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-LC13 Coughing. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.0115, Mixed Models Analysis; Mean Difference (Net) = -4.55, 95% CI 2-sided [-8.06 to -1.03]
Statistical Analysis 3: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-LC13 Haemoptysis. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.7824, Mixed Models Analysis; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.75 to 0.99]
Statistical Analysis 4: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-LC13 Sore Mouth. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.2988, Mixed Models Analysis; Mean Difference (Net) = 1.16, 95% CI 2-sided [-1.04 to 3.36]
Statistical Analysis 5: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-LC13 Dysphagia. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.1916, Mixed Models Analysis; Mean Difference (Net) = -1.51, 95% CI 2-sided [-3.79 to 0.76]
Statistical Analysis 6: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-LC13 Peripheral Neuropathy. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.0279, Mixed Models Analysis; Mean Difference (Net) = 5.37, 95% CI 2-sided [0.59 to 10.15]
Statistical Analysis 7: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-LC13 Alopecia. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.9162, Mixed Models Analysis; Mean Difference (Net) = -0.20, 95% CI 2-sided [-3.89 to 3.49]
Statistical Analysis 8: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-LC13 Pain in Chest. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.6698, Mixed Models Analysis; Mean Difference (Net) = -0.53, 95% CI 2-sided [-2.96 to 1.90]
Statistical Analysis 9: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-LC13 Pain in Arm or Shoulder. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.8035, Mixed Models Analysis; Mean Difference (Net) = 0.45, 95% CI 2-sided [-3.13 to 4.04]
Statistical Analysis 10: Comparison: Lorlatinib vs Crizotinib; This is the analysis for QLQ-LC13 Pain in Other Parts. Estimated change from baseline was based on random intercept random slope mixed-effects model with an intercept term, treatment, time (as a continuous variable), treatment-by-time, baseline and randomization stratification factors as covariates; Test type: Superiority; p = 0.1143, Mixed Models Analysis; Mean Difference (Net) = 3.36, 95% CI 2-sided [-0.82 to 7.55]

24. Secondary Outcome: Change From Baseline in Health Status as Assessed by EuroQol 5 Dimension 5 Level (EQ-5D-5L) - Visual Analogue Scale (VAS) Across Time
Description: The EuroQol EQ-5D-5L is a participant-completed questionnaire designed to assess health status. There are 2 components to the EuroQol EQ-5D-5L: a descriptive system in which individuals rate their level of problems (none, slight, moderate, severe, extreme/unable) in 5 areas (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a VAS. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state) and higher scores indicate better health state.
Time Frame: Baseline, Day 1 of all cycles from Cycle 2 to Cycle 38, and End of Treatment
Population: "Number of Participants Analyzed" included all participants in the EQ-5D-5L PRO analysis population within each treatment group. "Number Analyzed" included all participants with at least a baseline and postbaseline assessment at the visit.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 147 | 138
Units on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 143 | 133
  Cycle 2 Day 1 | 6.0 [3.33 to 8.72] | 3.1 [0.19 to 5.92]
  Cycle 3 Day 1: number analyzed (Participants) | 137 | 124
  Cycle 3 Day 1 | 6.0 [3.30 to 8.75] | 5.3 [2.37 to 8.18]
  Cycle 4 Day 1: number analyzed (Participants) | 133 | 122
  Cycle 4 Day 1 | 7.1 [3.71 to 10.41] | 5.6 [2.77 to 8.47]
  Cycle 5 Day 1: number analyzed (Participants) | 130 | 115
  Cycle 5 Day 1 | 4.3 [0.39 to 8.13] | 5.1 [1.88 to 8.26]
  Cycle 6 Day 1: number analyzed (Participants) | 127 | 105
  Cycle 6 Day 1 | 6.5 [3.11 to 9.85] | 4.5 [1.08 to 7.91]
  Cycle 7 Day 1: number analyzed (Participants) | 122 | 100
  Cycle 7 Day 1 | 5.5 [1.95 to 9.13] | 4.0 [0.35 to 7.55]
  Cycle 8 Day 1: number analyzed (Participants) | 125 | 94
  Cycle 8 Day 1 | 6.7 [2.95 to 10.37] | 4.2 [0.63 to 7.68]
  Cycle 9 Day 1: number analyzed (Participants) | 120 | 82
  Cycle 9 Day 1 | 6.4 [2.47 to 10.33] | 3.9 [0.09 to 7.69]
  Cycle 10 Day 1: number analyzed (Participants) | 116 | 74
  Cycle 10 Day 1 | 7.2 [3.22 to 11.20] | 3.9 [-0.02 to 7.75]
  Cycle 11 Day 1: number analyzed (Participants) | 117 | 73
  Cycle 11 Day 1 | 8.1 [4.27 to 11.83] | 2.0 [-1.62 to 5.59]
  Cycle 12 Day 1: number analyzed (Participants) | 117 | 61
  Cycle 12 Day 1 | 7.6 [3.82 to 11.41] | 4.8 [0.95 to 8.59]
  Cycle 13 Day 1: number analyzed (Participants) | 114 | 56
  Cycle 13 Day 1 | 7.5 [3.91 to 11.11] | 5.8 [1.99 to 9.51]
  Cycle 14 Day 1: number analyzed (Participants) | 110 | 48
  Cycle 14 Day 1 | 6.7 [3.06 to 10.32] | 2.3 [-1.33 to 5.91]
  Cycle 15 Day 1: number analyzed (Participants) | 111 | 43
  Cycle 15 Day 1 | 6.1 [2.33 to 9.96] | 1.5 [-3.14 to 6.07]
  Cycle 16 Day 1: number analyzed (Participants) | 104 | 39
  Cycle 16 Day 1 | 6.9 [2.71 to 11.04] | 2.4 [-2.89 to 7.71]
  Cycle 17 Day 1: number analyzed (Participants) | 93 | 32
  Cycle 17 Day 1 | 8.3 [4.08 to 12.46] | 1.1 [-5.05 to 7.17]
  Cycle 18 Day 1: number analyzed (Participants) | 83 | 29
  Cycle 18 Day 1 | 8.7 [4.17 to 13.28] | 1.3 [-5.01 to 7.56]
  Cycle 19 Day 1: number analyzed (Participants) | 78 | 23
  Cycle 19 Day 1 | 6.8 [1.86 to 11.70] | 2.8 [-2.79 to 8.44]
  Cycle 20 Day 1: number analyzed (Participants) | 69 | 19
  Cycle 20 Day 1 | 7.9 [2.83 to 13.06] | 3.4 [-3.59 to 10.44]
  Cycle 21 Day 1: number analyzed (Participants) | 65 | 17
  Cycle 21 Day 1 | 7.2 [1.96 to 12.44] | 3.3 [-4.06 to 10.64]
  Cycle 22 Day 1: number analyzed (Participants) | 56 | 14
  Cycle 22 Day 1 | 4.5 [-0.51 to 9.48] | 1.9 [-6.69 to 10.54]
  Cycle 23 Day 1: number analyzed (Participants) | 48 | 12
  Cycle 23 Day 1 | 5.2 [-0.68 to 11.14] | -0.6 [-10.97 to 9.81]
  Cycle 24 Day 1: number analyzed (Participants) | 44 | 10
  Cycle 24 Day 1 | 4.9 [-1.22 to 11.09] | -3.0 [-21.43 to 15.43]
  Cycle 25 Day 1: number analyzed (Participants) | 39 | 9
  Cycle 25 Day 1 | 4.0 [-2.13 to 10.18] | 1.4 [-11.86 to 14.75]
  Cycle 26 Day 1: number analyzed (Participants) | 35 | 9
  Cycle 26 Day 1 | 7.9 [1.00 to 14.77] | 2.0 [-11.84 to 15.84]
  Cycle 27 Day 1: number analyzed (Participants) | 30 | 7
  Cycle 27 Day 1 | 4.6 [-2.37 to 11.57] | 3.0 [-12.79 to 18.79]
  Cycle 28 Day 1: number analyzed (Participants) | 23 | 6
  Cycle 28 Day 1 | 6.0 [-3.75 to 15.66] | 2.7 [-13.20 to 18.54]
  Cycle 29Day 1: number analyzed (Participants) | 20 | 5
  Cycle 29Day 1 | 7.4 [-3.78 to 18.48] | 8.2 [-11.18 to 27.58]
  Cycle 30 Day 1: number analyzed (Participants) | 14 | 4
  Cycle 30 Day 1 | 9.1 [-5.66 to 23.95] | 2.8 [-22.92 to 28.42]
  Cycle 31 Day 1: number analyzed (Participants) | 12 | 2
  Cycle 31 Day 1 | 7.8 [-11.84 to 27.51] | 0.0 [-190.59 to 190.59]
  Cycle 32 Day 1: number analyzed (Participants) | 10 | 2
  Cycle 32 Day 1 | 7.9 [-11.65 to 27.45] | 2.5 [-156.33 to 161.33]
  Cycle 33 Day 1: number analyzed (Participants) | 8 | 2
  Cycle 33 Day 1 | 4.4 [-21.74 to 30.49] | -2.5 [-224.86 to 219.86]
  Cycle 34 Day 1: number analyzed (Participants) | 6 | 1
  Cycle 34 Day 1 | -0.5 [-32.20 to 31.20] | 20.0
  Cycle 35 Day 1: number analyzed (Participants) | 4 | 1
  Cycle 35 Day 1 | 0.0 [-32.48 to 32.48] | 20.0
  Cycle 36 Day 1: number analyzed (Participants) | 2 | 1
  Cycle 36 Day 1 | -4.5 [-315.80 to 306.80] | 15.0
  Cycle 37 Day 1: number analyzed (Participants) | 2 | 0
  Cycle 37 Day 1 | -17.5 [-176.33 to 141.33] |
  Cycle 38 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 38 Day 1 | 25.0 |
  End of Treatment: number analyzed (Participants) | 27 | 82
  End of Treatment | -3.7 [-13.66 to 6.33] | -1.3 [-5.43 to 2.80]

25. Secondary Outcome: Change From Baseline in Health Status as Assessed by EuroQol 5 Dimension 5 Level (EQ-5D-5L) - Index Across Time
Description: The EuroQol EQ-5D-5L is a participant-completed questionnaire designed to assess health status. There are 2 components to the EuroQol EQ-5D-5L: a descriptive system in which individuals rate their level of problems (none, slight, moderate, severe, extreme/unable) in 5 areas (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a VAS in which participants rate their overall health status from 0 (worst imaginable) to 100 (best imaginable). EQ-5D summary index is obtained with a formula that weights each level of the 5 dimensions. The index-based score is interpreted along a continuum of 0 (death) to 1 (perfect health).
Time Frame: Baseline, Day 1 of all cycles from Cycle 2 to Cycle 38, and End of Treatment
Population: "Number of Participants Analyzed" included all participants in the PRO analysis population within each treatment group. "Number Analyzed" included all participants with at least a baseline and postbaseline assessment at the visit.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 148 | 140
Units on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 141 | 133
  Cycle 2 Day 1 | 0.078 [0.0475 to 0.1092] | 0.064 [0.0258 to 0.1021]
  Cycle 3 Day 1: number analyzed (Participants) | 138 | 124
  Cycle 3 Day 1 | 0.071 [0.0327 to 0.1097] | 0.101 [0.0665 to 0.1353]
  Cycle 4 Day 1: number analyzed (Participants) | 131 | 121
  Cycle 4 Day 1 | 0.089 [0.0520 to 0.1254] | 0.098 [0.0619 to 0.1338]
  Cycle 5 Day 1: number analyzed (Participants) | 130 | 114
  Cycle 5 Day 1 | 0.047 [0.0061 to 0.0887] | 0.100 [0.0626 to 0.1373]
  Cycle 6 Day 1: number analyzed (Participants) | 126 | 104
  Cycle 6 Day 1 | 0.077 [0.0407 to 0.1124] | 0.070 [0.0324 to 0.1077]
  Cycle 7 Day 1: number analyzed (Participants) | 121 | 99
  Cycle 7 Day 1 | 0.062 [0.0180 to 0.1052] | 0.046 [0.0002 to 0.0910]
  Cycle 8 Day 1: number analyzed (Participants) | 124 | 93
  Cycle 8 Day 1 | 0.074 [0.0340 to 0.1133] | 0.061 [0.0201 to 0.1011]
  Cycle 9 Day 1: number analyzed (Participants) | 118 | 82
  Cycle 9 Day 1 | 0.060 [0.0175 to 0.1028] | 0.050 [0.0082 to 0.0919]
  Cycle 10 Day 1: number analyzed (Participants) | 115 | 75
  Cycle 10 Day 1 | 0.074 [0.0303 to 0.1179] | 0.050 [0.0168 to 0.0826]
  Cycle 11 Day 1: number analyzed (Participants) | 116 | 73
  Cycle 11 Day 1 | 0.083 [0.0418 to 0.1237] | 0.057 [0.0222 to 0.0914]
  Cycle 12 Day 1: number analyzed (Participants) | 116 | 61
  Cycle 12 Day 1 | 0.080 [0.0390 to 0.1201] | 0.049 [0.0118 to 0.0864]
  Cycle 13 Day 1: number analyzed (Participants) | 113 | 56
  Cycle 13 Day 1 | 0.081 [0.0365 to 0.1259] | 0.055 [0.0165 to 0.0931]
  Cycle 14 Day 1: number analyzed (Participants) | 110 | 48
  Cycle 14 Day 1 | 0.091 [0.0490 to 0.1322] | 0.021 [-0.0157 to 0.0576]
  Cycle 15 Day 1: number analyzed (Participants) | 110 | 43
  Cycle 15 Day 1 | 0.077 [0.0314 to 0.1217] | 0.036 [-0.0100 to 0.0811]
  Cycle 16 Day 1: number analyzed (Participants) | 103 | 39
  Cycle 16 Day 1 | 0.091 [0.0469 to 0.1347] | 0.051 [0.0070 to 0.0953]
  Cycle 17 Day 1: number analyzed (Participants) | 91 | 31
  Cycle 17 Day 1 | 0.098 [0.0523 to 0.1434] | -0.016 [-0.1000 to 0.0685]
  Cycle 18 Day 1: number analyzed (Participants) | 84 | 28
  Cycle 18 Day 1 | 0.103 [0.0520 to 0.1531] | 0.021 [-0.0296 to 0.0716]
  Cycle 19 Day 1: number analyzed (Participants) | 79 | 21
  Cycle 19 Day 1 | 0.100 [0.0481 to 0.1518] | 0.027 [-0.0246 to 0.0793]
  Cycle 20 Day 1: number analyzed (Participants) | 69 | 18
  Cycle 20 Day 1 | 0.103 [0.0459 to 0.1596] | 0.025 [-0.0593 to 0.1090]
  Cycle 21 Day 1: number analyzed (Participants) | 65 | 17
  Cycle 21 Day 1 | 0.068 [0.0091 to 0.1276] | 0.040 [-0.0187 to 0.0989]
  Cycle 22 Day 1: number analyzed (Participants) | 56 | 14
  Cycle 22 Day 1 | 0.079 [0.0134 to 0.1447] | 0.052 [-0.0249 to 0.1289]
  Cycle 23 Day 1: number analyzed (Participants) | 48 | 12
  Cycle 23 Day 1 | 0.060 [-0.0127 to 0.1324] | 0.006 [-0.2020 to 0.2133]
  Cycle 24 Day 1: number analyzed (Participants) | 44 | 10
  Cycle 24 Day 1 | 0.082 [0.0104 to 0.1531] | -0.053 [-0.2793 to 0.1731]
  Cycle 25 Day 1: number analyzed (Participants) | 39 | 9
  Cycle 25 Day 1 | 0.047 [-0.0287 to 0.1231] | 0.045 [-0.0289 to 0.1194]
  Cycle 26 Day 1: number analyzed (Participants) | 35 | 9
  Cycle 26 Day 1 | 0.065 [-0.0218 to 0.1519] | 0.039 [-0.0200 to 0.0978]
  Cycle 27 Day 1: number analyzed (Participants) | 30 | 7
  Cycle 27 Day 1 | 0.042 [-0.0603 to 0.1434] | 0.021 [-0.0867 to 0.1292]
  Cycle 28 Day 1: number analyzed (Participants) | 23 | 6
  Cycle 28 Day 1 | 0.024 [-0.0911 to 0.1399] | -0.040 [-0.1640 to 0.0836]
  Cycle 29 Day 1: number analyzed (Participants) | 20 | 5
  Cycle 29 Day 1 | 0.046 [-0.0836 to 0.1755] | 0.041 [-0.0108 to 0.0928]
  Cycle 30 Day 1: number analyzed (Participants) | 14 | 4
  Cycle 30 Day 1 | 0.099 [-0.0355 to 0.2306] | -0.028 [-0.1740 to 0.1190]
  Cycle 31 Day 1: number analyzed (Participants) | 12 | 2
  Cycle 31 Day 1 | 0.086 [-0.0957 to 0.2683] | -0.024 [-0.8558 to 0.8088]
  Cycle 32 Day 1: number analyzed (Participants) | 10 | 2
  Cycle 32 Day 1 | 0.058 [-0.1601 to 0.2767] | -0.139 [-2.4320 to 2.1550]
  Cycle 33 Day 1: number analyzed (Participants) | 8 | 2
  Cycle 33 Day 1 | 0.058 [-0.2006 to 0.3163] | -0.024 [-0.8558 to 0.8088]
  Cycle 34 Day 1: number analyzed (Participants) | 6 | 1
  Cycle 34 Day 1 | 0.062 [-0.2820 to 0.4057] | 0.042
  Cycle 35 Day 1: number analyzed (Participants) | 4 | 1
  Cycle 35 Day 1 | 0.129 [-0.1098 to 0.3668] | 0.042
  Cycle 36 Day 1: number analyzed (Participants) | 2 | 1
  Cycle 36 Day 1 | -0.027 [-1.7736 to 1.7206] | 0.042
  Cycle 37 Day 1: number analyzed (Participants) | 2 | 0
  Cycle 37 Day 1 | 0.056 [-0.6497 to 0.7607] |
  Cycle 38 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 38 Day 1 | 0.232 |
  End of Treatment: number analyzed (Participants) | 27 | 79
  End of Treatment | -0.033 [-0.1513 to 0.0852] | 0.001 [-0.0769 to 0.0782]

26. Secondary Outcome: Time to Deterioration (TTD) in Participant Reported Pain in Chest, Dyspnea, or Cough From QLQ-LC13
Description: The EORTC QLQ LC13 consists of 13 questions and includes 1 multi-item scale and 9 single items assessing symptoms (dyspnea, cough, haemoptysis, and site-specific pain), side effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia), and pain medication use. The scale scores rang from 0 to 100, with higher scores indicating higher ("worse") level of symptoms. TTD in pain in chest, dyspnea, or cough was defined as the time from randomization to the first time the participant's score showed a 10 point or greater increase after baseline in any of the 3 symptoms. TTD in months was calculated as (date of deterioration or censoring - randomization date +1)/30.4375.
Time Frame: From Baseline up to 33 months
Population: Participants in the EORTC QLQ-LC13 PRO analysis population with change from baseline scores within each treatment group and subscale.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 146 | 139
Months | 3.3 [2.1 to 4.7] | 3.7 [2.0 to 5.5]
Statistical Analysis 1: Comparison: Lorlatinib vs Crizotinib; Test type: Superiority; p = 0.7293, one-sided stratified log-rank; Stratified by the presence of brain metastases (Yes/No) and ethnic origin (Asian/Non-Asian) at randomization; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.822 to 1.444] — [estimate comment as in outcome 1, analysis 1]

27. Secondary Outcome: Number of Participant With ALK Domain Mutation in Plasma Circulating Nucleic Acid (CNA) Analysis at Screening, Cycle 2 Day 1 and Cycle 7 Day 1
Description: The analysis of anaplastic lymphoma kinase (ALK) domain mutation in plasma CNA was performed by next-generation sequencing (NGS) and the number of participants with one or more ALK mutations at Screening, Cycle 2 Day 1 and Cycle 7 Day 1 is presented here.
Time Frame: at Screening, Cycle 2 Day 1 and Cycle 7 Day 1
Population: "Number of Participants Analyzed" included all participants in the plasma CNA analysis population within each treatment group at screening. "Number Analyzed" included all participants in the plasma CNA analysis population within each treatment group at the specified visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 130 | 125
Participants
  at Screening: ≥1 ALK Mutation Detected | 5 | 6
  at Screening: No ALK Mutation Detected | 88 | 91
  at Screening: No Circulating Free Deoxyribonucleic Acid (cfDNA) Detected | 32 | 25
  at Screening: Other (Sample failed analysis, uninformative, or not analyzed.) | 5 | 3
  Cycle 2 Day 1: number analyzed (Participants) | 125 | 118
  Cycle 2 Day 1: ≥1 ALK Mutation Detected | 2 | 3
  Cycle 2 Day 1: No ALK Mutation Detected | 66 | 55
  Cycle 2 Day 1: No Circulating Free Deoxyribonucleic Acid (cfDNA) Detected | 53 | 58
  Cycle 2 Day 1: Other (Sample failed analysis, uninformative, or not analyzed.) | 4 | 2
  Cycle 7 Day 1: number analyzed (Participants) | 103 | 84
  Cycle 7 Day 1: ≥1 ALK Mutation Detected | 3 | 5
  Cycle 7 Day 1: No ALK Mutation Detected | 45 | 42
  Cycle 7 Day 1: No Circulating Free Deoxyribonucleic Acid (cfDNA) Detected | 52 | 35
  Cycle 7 Day 1: Other (Sample failed analysis, uninformative, or not analyzed.) | 3 | 2

28. Secondary Outcome: Number of Participant With ALK Fusion Variant in Plasma Circulating Nucleic Acid (CNA) Analysis at Screening, Cycle 2 Day 1 and Cycle 7 Day 1
Description: The analysis of ALK fusion variant in plasma CNA was performed by NGS and the number of participants with fusion variants at Screening, Cycle 2 Day 1 and Cycle 7 Day 1 is presented here. In the table below, EML4-ALK is the abbreviation of echinoderm microtubule-associated protein-like 4 anaplastic lymphoma kinase.
Time Frame: at Screening, Cycle 2 Day 1 and Cycle 7 Day 1
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib | Crizotinib
Number analyzed (Participants) | 130 | 125
Participants
  at Screening: EML4-ALK Variant 1 | 19 | 25
  at Screening: EML4-ALK Variant 2 | 7 | 2
  at Screening: EML4-ALK Variant 3 | 18 | 21
  at Screening: EML4-ALK Other | 15 | 9
  at Screening: ALK Rearrangement Other | 2 | 4
  at Screening: ALK Rearrangement Not Detected | 32 | 36
  at Screening: No cfDNA Detected | 32 | 25
  at Screening: Other (Sample failed analysis, uninformative, or not analyzed.) | 5 | 3
  Cycle 2 Day 1: number analyzed (Participants) | 125 | 118
  Cycle 2 Day 1: EML4-ALK Variant 1 | 1 | 7
  Cycle 2 Day 1: EML4-ALK Variant 2 | 2 | 0
  Cycle 2 Day 1: EML4-ALK Variant 3 | 2 | 2
  Cycle 2 Day 1: EML4-ALK Other | 2 | 1
  Cycle 2 Day 1: ALK Rearrangement Other | 0 | 0
  Cycle 2 Day 1: ALK Rearrangement Not Detected | 61 | 48
  Cycle 2 Day 1: No cfDNA Detected | 53 | 58
  Cycle 2 Day 1: Other (Sample failed analysis, uninformative, or not analyzed.) | 4 | 2
  Cycle 7 Day 1: number analyzed (Participants) | 103 | 84
  Cycle 7 Day 1: EML4-ALK Variant 1 | 0 | 5
  Cycle 7 Day 1: EML4-ALK Variant 2 | 0 | 1
  Cycle 7 Day 1: EML4-ALK Variant 3 | 0 | 4
  Cycle 7 Day 1: EML4-ALK Other | 0 | 1
  Cycle 7 Day 1: ALK Rearrangement Other | 0 | 2
  Cycle 7 Day 1: ALK Rearrangement Not Detected | 48 | 34
  Cycle 7 Day 1: No cfDNA Detected | 52 | 35
  Cycle 7 Day 1: Other (Sample failed analysis, uninformative, or not analyzed.) | 3 | 2

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment through end of study follow-up (infinite lag) or start of new anti-cancer therapy, whichever occurred first (assessed up to 33 months).
Description: The analysis of adverse events included all participants who received at least 1 dose of study drug. Participants were classified according to the treatment assigned at randomization. Totals number of participants at a higher level were not necessarily the sum of those at the lower levels since a participant may report two or more different adverse events within the higher level category.
Arm/Group | Lorlatinib | Crizotinib
All-Cause Mortality (participants affected / at risk) | 23/149 | 28/142
Serious Adverse Events (participants affected / at risk) | 51/149 | 39/142
Other Adverse Events (participants affected / at risk) | 148/149 | 140/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lorlatinib (N=149) | Crizotinib (N=142)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Blindness cortical (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 1
Disease progression (General disorders) | 1 | 1
Generalised oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 3
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Haemophilus infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 5
Pneumonia cryptococcal (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Follicle centre lymphoma, follicular grade I, II, III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 1 | 0
Thalamus haemorrhage (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract disorder (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Radiotherapy to bone (Surgical and medical procedures) | 1 | 0
Aortitis (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lorlatinib (N=149) | Crizotinib (N=142)
Anaemia (Blood and lymphatic system disorders) | 29 | 11
Neutropenia (Blood and lymphatic system disorders) | 10 | 21
Bradycardia (Cardiac disorders) | 2 | 17
Sinus bradycardia (Cardiac disorders) | 4 | 15
Tinnitus (Ear and labyrinth disorders) | 9 | 1
Photopsia (Eye disorders) | 1 | 24
Vision blurred (Eye disorders) | 11 | 4
Visual impairment (Eye disorders) | 10 | 16
Abdominal distension (Gastrointestinal disorders) | 9 | 3
Abdominal pain (Gastrointestinal disorders) | 7 | 11
Constipation (Gastrointestinal disorders) | 26 | 41
Diarrhoea (Gastrointestinal disorders) | 32 | 74
Flatulence (Gastrointestinal disorders) | 11 | 3
Nausea (Gastrointestinal disorders) | 22 | 74
Vomiting (Gastrointestinal disorders) | 19 | 55
Asthenia (General disorders) | 20 | 27
Chest pain (General disorders) | 16 | 20
Fatigue (General disorders) | 11 | 24
Oedema (General disorders) | 16 | 13
Oedema peripheral (General disorders) | 65 | 44
Pain (General disorders) | 5 | 8
Pyrexia (General disorders) | 22 | 16
Bronchitis (Infections and infestations) | 9 | 3
Nasopharyngitis (Infections and infestations) | 8 | 10
Pneumonia (Infections and infestations) | 5 | 8
Respiratory tract infection (Infections and infestations) | 12 | 6
Upper respiratory tract infection (Infections and infestations) | 16 | 11
Urinary tract infection (Infections and infestations) | 6 | 10
Alanine aminotransferase increased (Investigations) | 26 | 48
Amylase increased (Investigations) | 13 | 16
Aspartate aminotransferase increased (Investigations) | 21 | 39
Blood alkaline phosphatase increased (Investigations) | 7 | 18
Blood cholesterol increased (Investigations) | 59 | 4
Blood creatine phosphokinase increased (Investigations) | 16 | 24
Blood creatinine increased (Investigations) | 9 | 19
Blood lactate dehydrogenase increased (Investigations) | 3 | 15
Blood triglycerides increased (Investigations) | 19 | 2
Electrocardiogram QT prolonged (Investigations) | 5 | 8
Gamma-glutamyltransferase increased (Investigations) | 22 | 22
Lipase increased (Investigations) | 14 | 17
Neutrophil count decreased (Investigations) | 3 | 16
Weight decreased (Investigations) | 4 | 10
Weight increased (Investigations) | 57 | 18
White blood cell count decreased (Investigations) | 1 | 11
Decreased appetite (Metabolism and nutrition disorders) | 5 | 35
Dyslipidaemia (Metabolism and nutrition disorders) | 9 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 53 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 5
Hyperlipidaemia (Metabolism and nutrition disorders) | 16 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 78 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 12 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 18
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 16
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 | 12
Dizziness (Nervous system disorders) | 16 | 20
Dysgeusia (Nervous system disorders) | 8 | 23
Headache (Nervous system disorders) | 25 | 25
Hypoaesthesia (Nervous system disorders) | 8 | 7
Memory impairment (Nervous system disorders) | 13 | 3
Neuropathy peripheral (Nervous system disorders) | 13 | 0
Paraesthesia (Nervous system disorders) | 18 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 1
Anxiety (Psychiatric disorders) | 10 | 3
Insomnia (Psychiatric disorders) | 14 | 13
Proteinuria (Renal and urinary disorders) | 9 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 26
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 23
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 | 0
Rash (Skin and subcutaneous tissue disorders) | 15 | 11
Hypertension (Vascular disorders) | 27 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT03052608/Prot_001.pdf
  • Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT03052608/SAP_000.pdf